CLINICAL TRIAL: NCT04857437
Title: A PHASE 1, 3-PART, SPONSOR OPEN STUDY OF PF-07202954 IN HEALTHY ADULTS: RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TO ASSESS SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE (IN PART 1), AND REPEATED (IN PART 2), ESCALATING, ORAL DOSES ALONG WITH CONDITIONAL PART 3 OF RANDOMIZED, OPEN-LABEL ASSESSMENT OF EFFECT OF FOOD ON PF-07202954 EXPOSURE
Brief Title: Study in Healthy Adults Evaluating PF-07202954
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4171001; 2020-002121-28 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Single, Escalating Doses of PF-07202954 or Placebo (Cohorts 1 and 2)
  Interventions: Drug: PF-07202954 Single Dose; Drug: Placebo
- Part 2 (Experimental): Repeated, Escalating Doses of PF-07202954 or placebo from Day 1 to Day 14, inclusive (Cohorts 3, 4, 5, 6 7, and optional Cohort 8)
  Interventions: Drug: PF-07202954 Repeat Dose; Drug: Placebo
- Part 3 (Experimental): Single dose of PF-07202954 with a high-fat/high-caloric meal and a single dose following an overnight fast of ≥10 hours
  Interventions: Drug: PF-07202954 Single Dose

INTERVENTIONS:
Drug: PF-07202954 Repeat Dose — 10, 30, 100, 300, 600, 1200 milligrams (mg)
  Arms: Part 2
Drug: PF-07202954 Single Dose — 10, 30, 100, 300, 600, 900, 1200 milligrams (mg)
  Arms: Part 1; Part 3
Drug: Placebo — Matching Placebo
  Arms: Part 1; Part 2

SUMMARY:
The study is planned as a 3 part design with investigator and participant blinded (sponsor-open), placebo controlled, randomized, dose escalation in Part 1 and Part 2; and a randomized, open label design, in Part 3 (if conducted).

ELIGIBILITY:
Inclusion Criteria:- healthy subjects (all 3 Parts)

* evidence of steatosis on FibroScan (Part 2 only)
* BMI 17.5 to 30.5 kg/m2 (Part 1, Part 3)
* BMI 17.5 to 35.4 kg/m2 (Part 2) Exclusion Criteria:- evidence of clinically significant disease
* subjects on chronic medications
* clinically significant, abnormal laboratory results, vital signs, or cardiac conduction abnormalities
* contraindication to MRI (Part 2, only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4171001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study originally had 3 parts. Sponsor strategically decided not to conduct Part 2 and 3, based on results from Part 1 of the study. This decision was not due to any safety concern from Part 1 of the study. The study was concluded following Part 1; hence, no participants were enrolled in Part 2 and 3.
Groups:
- Part1 Cohort1: Placebo/PF-07202954 100mg Std Meal/PF-07202954 600mg/PF-07202954 100mg High Fat Meal: Participants were administered a single oral dose of placebo with a standard (std) meal on Day 1 of Period 1 followed by a single oral dose of PF-07202954 100 mg with a std meal on Day 1 of Period 2. Participants received a single oral dose of PF-07202954 600 mg with a std meal and PF-07202954 100 mg with high fat/high calorie meal on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort1: PF-07202954 10mg/Placebo/PF-07202954 600mg/PF-07202954 100mg High Fat Meal: Participants were administered a single oral dose of PF-07202954 10 mg with a std meal on Day 1 of Period 1 followed by a single oral dose of placebo with a std meal on Day 1 of Period 2. Participants received a single oral dose of PF-07202954 600 mg with a std meal and PF-07202954 100 mg with high fat/high calorie meal on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/Placebo/PF-07202954 100mg High Fat Meal: Participants were administered a single oral dose of PF-07202954 10 mg with a std meal on Day 1 of Period 1 followed by a single oral dose of PF-07202954 100 mg with a std meal on Day 1 of Period 2. Participants received a single oral dose of placebo with a std meal and PF-07202954 100 mg with high fat/high calorie meal on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/PF-07202954 600mg/Placebo: Participants were administered a single oral dose of PF-07202954 10 mg with a std meal on Day 1 of Period 1 followed by a single oral dose of PF-07202954 100 mg with a std meal on Day 1 of Period 2. Participants received a single oral dose of PF-07202954 600 mg and placebo with std meal on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort2: Placebo/PF-07202954 300mg/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted: Participants were administered a single oral dose of placebo with a std meal on Day 1 of Period 1 followed by a single oral dose of PF-07202954 300 mg with a std meal on Day 1 of Period 2. Participants received a single oral dose of PF-07202954 100 mg with a std meal and PF-07202954 100 mg under fasting condition on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort2: PF-07202954 30mg/Placebo/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted: Participants were administered a single oral dose of PF-07202954 30 mg with a std meal on Day 1 of Period 1 followed by a single oral dose of placebo with a std meal on Day 1 of Period 2. Participants received a single oral dose of PF-07202954 100 mg with a std meal and PF-07202954 100 mg under fasting condition on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/Placebo/PF-07202954 100mg Fasted: Participants were administered a single oral dose of PF-07202954 30 mg with a std meal on Day 1 of Period 1 followed by a single oral dose of PF-07202954 300 mg with a std meal on Day 1 of Period 2. Participants received a single oral dose of placebo with a std meal and PF-07202954 100 mg under fasting condition on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
- Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/PF-07202954 100mg Std Meal/Placebo: Participants were administered a single oral dose of PF-07202954 30 mg with a std meal on Day 1 of Period 1 followed by a single oral dose of PF-07202954 300 mg with a std meal on Day 1 of Period 2. Participants received a single oral dose of PF-07202954 100 mg and placebo with a std meal on Day 1 of Periods 3 and 4, respectively. The dosing in each period was separated by an interval of at least 10 days. Participants were followed up for approximately 28 days after last dose of study treatment in Period 4.
Period: Part 1 Period 1
Arm/Group | Part1 Cohort1: Placebo/PF-07202954 100mg Std Meal/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/Placebo/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/Placebo/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/PF-07202954 600mg/Placebo | Part1 Cohort2: Placebo/PF-07202954 300mg/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/Placebo/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/Placebo/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/PF-07202954 100mg Std Meal/Placebo
Started | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 2
Arm/Group | Part1 Cohort1: Placebo/PF-07202954 100mg Std Meal/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/Placebo/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/Placebo/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/PF-07202954 600mg/Placebo | Part1 Cohort2: Placebo/PF-07202954 300mg/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/Placebo/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/Placebo/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/PF-07202954 100mg Std Meal/Placebo
Started | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 3
Arm/Group | Part1 Cohort1: Placebo/PF-07202954 100mg Std Meal/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/Placebo/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/Placebo/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/PF-07202954 600mg/Placebo | Part1 Cohort2: Placebo/PF-07202954 300mg/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/Placebo/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/Placebo/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/PF-07202954 100mg Std Meal/Placebo
Started | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1 (One participant did not enter Period 3 as participant was unable to return to unit)
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 4
Arm/Group | Part1 Cohort1: Placebo/PF-07202954 100mg Std Meal/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/Placebo/PF-07202954 600mg/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/Placebo/PF-07202954 100mg High Fat Meal | Part1 Cohort1: PF-07202954 10mg/PF-07202954 100mg Std Meal/PF-07202954 600mg/Placebo | Part1 Cohort2: Placebo/PF-07202954 300mg/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/Placebo/PF-07202954 100mg Std Meal/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/Placebo/PF-07202954 100mg Fasted | Part1 Cohort2: PF-07202954 30mg/PF-07202954 300mg/PF-07202954 100mg Std Meal/Placebo
Started | 2 | 1 | 2 | 1 | 2 | 0 (Participant withdrawn prior to dosing as eligibility criteria was no longer met.) | 0 (Participant withdrawn prior to dosing as eligibility criteria was no longer met.) | 1
Completed | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data has been presented for all participants in Cohort 1 and 2 as presenting the data per sequence would risk re-identification of participants due to low enrollment of participants per sequence. The study was concluded following Part 1; hence, no participants were enrolled in Part 2 and 3.
Groups:
- Part 1 Cohort 1: All Participants: All participants who were randomized to either of the four treatment sequences in Cohort 1 and received placebo and escalating doses of PF-07202954 either with std meal or with high fat/high calorie meal in Periods 1, 2, 3 or 4 were included. All doses were administered once on Day 1 of each period via the oral route. The dosing in each period was separated by an interval of at least 10 days.
- Part 1 Cohort 2: All Participants: All participants who were randomized to either of the four treatment sequences in Cohort 2 and received placebo and escalating doses of PF-07202954 with either std meal or under fasting condition in Period 1, 2, 3 or 4 were included. All doses were administered once on Day 1 of each period via the oral route. The dosing in each period was separated by an interval of at least 10 days.
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: All Participants | Part 1 Cohort 2: All Participants | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were AEs that occurred following the start of study treatment (either PF-07202954 or placebo) up to approximately 28 days after the last dose.
Time Frame: From start of study treatment on Day 1 up to 28 days post last dose of study treatment (maximum up to 10 weeks)
Population: Safety population included all participants who were randomly assigned to study treatment and who took at least 1 dose of study treatment. Treatment groups with same dose and administration were combined as planned.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 and 2: Placebo: Part 1: Participants were administered a single oral dose of placebo with a standard meal on Day 1 of any treatment period.
- Cohort 1: PF-07202954 10 mg: Part 1: Participants were administered a single oral dose of PF-07202954 10 mg with a standard meal on Day 1 of any treatment period.
- Cohort 2: PF-07202954 30 mg: Part 1: Participants were administered a single oral dose of PF-07202954 30 mg with a standard meal on Day 1 of any treatment period.
- Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1: Participants were administered a single oral dose of PF-07202954 100 mg with a standard meal on Day 1 of any treatment period.
- Cohort 2: PF-07202954 300 mg: Part 1: Participants were administered a single oral dose of PF-07202954 300 mg with a standard meal on Day 1 of any treatment period.
- Cohort 1: PF-07202954 600 mg: Part 1: Participants were administered a single oral dose of PF-07202954 600 mg with a standard meal on Day 1 of any treatment period.
- Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1: Participants were administered a single oral dose of PF-07202954 100 mg with a high fat/ high calorie meal on Day 1 of any treatment period.
- Cohort 2: PF-07202954 100 mg Fasted: Part 1: Participants were administered a single oral dose of PF-07202954 100 mg under fasting condition on Day 1 of any treatment period.
Arm/Group | Cohort 1 and 2: Placebo: Part 1 | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 11 | 4 | 4 | 9 | 5 | 4 | 5 | 2
Participants | 3 | 0 | 1 | 2 | 1 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Laboratory Abnormalities Meeting Pre-defined Criteria: Part 1
Description: Pre-defined criteria for laboratory abnormalities included, hematology: neutrophils/leukocytes (less than [<] 0.8* lower limit normal [LLN]); monocytes/leukocytes (greater than [>] 1.2* upper limit normal [ULN]); clinical chemistry: low density lipoprotein (LDL) (>1.2*ULN), creatine kinase (>2.0*ULN); and urinalysis: specific gravity (<1.003); ketones, urine protein, urine hemoglobin, nitrite (greater than equal to [>=1]), urine erythrocytes (>= 20), red blood cells (RBC) casts (>1), bacteria (>20). Number of participants with any laboratory abnormality meeting pre-defined criteria was reported in this outcome measure.
Time Frame: From start of study treatment on Day 1 up to 28 days post last dose of study treatment (maximum up to 10 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo: Part 1 | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 11 | 4 | 4 | 9 | 5 | 4 | 5 | 2
Participants | 0 | 2 | 3 | 6 | 5 | 3 | 4 | 2

3. Primary Outcome: Number of Participants According to Categorization of Vital Signs Data: Part 1
Description: Vital signs were categorized according to the following criteria for potential clinical concern: diastolic blood pressure (DBP): <50 millimeter of mercury (mmHg), increase from baseline >= 20mmHg; systolic blood pressure (SBP): <90 mmHg, increase from baseline >=30mmHg; pulse rate: <40 beats per minute (bpm), >120 bpm.
Time Frame: From start of study treatment on Day 1 up to 28 days post last dose of study treatment (maximum up to 10 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo: Part 1 | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 11 | 4 | 4 | 9 | 5 | 4 | 5 | 2
Participants
  DBP: <50 mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  DBP: Increase from baseline >=20mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: <90 mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SBP: Increase from baseline >=30 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate: <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate: >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants According to Categorization of Electrocardiogram (ECG) Data: Part 1
Description: ECG parameters were categorized according to the following criteria for potential clinical concern: PR interval aggregate (msec) >=300, percent change >=25/50 percent (%); QRS duration, aggregate (msec) >=140, percent change >= 50%; QT interval corrected by Fridericia's formula (QTcF) interval aggregate (msec): >450 to <=480, > 480 to <=500, >500, change from baseline: >30 to <=60 and change >60.
Time Frame: From start of study treatment on Day 1 up to 28 days post last dose of study treatment (maximum up to 10 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: Placebo: Part 1 | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 11 | 4 | 4 | 9 | 5 | 4 | 5 | 2
Participants
  PR interval aggregate (msec): >=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval aggregate (msec): percent change >=25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration, aggregate (msec): >=140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration, aggregate (msec): percent change >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (msec): >450 to <=480 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (msec): >480 to <=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (msec): >=500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (msec): >30 to <=60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF interval aggregate (msec): change >60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs: Part 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to a maximum of 12 weeks
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Groups:
- Placebo: Part 2: Participants were planned to receive once daily oral dose of PF-07202954 matching placebo with a standard meal for 14 days.
- PF-07202954: Part 2: Participants were planned to receive once daily escalating oral doses of PF-07202954 with a standard meal for 14 days.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities Meeting Pre-defined Criteria: Part 2
Description: Pre-defined criteria for laboratory abnormalities included, hematology: neutrophils/leukocytes (<0.8* LLN); monocytes/leukocytes (>1.2* ULN); clinical chemistry: LDL (>1.2*ULN), creatine kinase (>2.0*ULN); and urinalysis: specific gravity (<1.003); ketones, urine protein, urine hemoglobin, nitrite (>=1), urine erythrocytes (>=20), RBC casts (>1), bacteria (>20).
Time Frame: Up to a maximum of 12 weeks
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Number of Participants According to Categorization of Vital Signs Data: Part 2
Description: Vital signs were planned to be categorized according to the following criteria for potential clinical concern: diastolic blood pressure: <50 mmHg, increase from baseline >=20mmHg; systolic blood pressure: <90 mmHg, increase from baseline >=30mmHg; pulse rate: <40 bpm, >120 bpm.
Time Frame: Up to a maximum of 12 weeks
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Number of Participants According to Categorization of ECG Data: Part 2
Description: ECG parameters were planned to be categorized according to the following criteria for potential clinical concern: PR interval aggregate (msec) >=300, percent change >=25/50%; QRS duration, aggregate (msec) >=140, percent change >=50%; QTcF interval aggregate (msec): >450 to <=480, >480 to <=500, >500, change from baseline: >30 to <=60 and change >60.
Time Frame: Up to a maximum of 12 weeks
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07202954: Part 3
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Groups:
- PF-07202954 With High-fat/High-calorie Meal: Part 3: Participants were planned to receive a single oral dose of PF-07202954 with high-fat/high-calorie meal in either Period 1 or 2.
- PF-07202954 Without High-fat/High-calorie Meal: Part 3: Participants were planned to receive a single oral dose of PF-07202954 without high-fat/high-calorie meal in either Period 1 or 2.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Time for Cmax (Tmax) of PF-07202954: Part 3
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Groups:
- PF-07202954 High-fat/High-caloric Meal: Part 3: Participants were planned to randomize to receive PF-07202954 with high-fat/high-caloric meal. Participants were planned to be followed up to 32 days.
- PF-07202954 Without High-fat/High-caloric Meal: Part 3: Participants were planned to randomize to receive PF-07202954 without high-fat/high-caloric meal. Participants were planned to be followed up to 32 days.
Arm/Group | PF-07202954 High-fat/High-caloric Meal: Part 3 | PF-07202954 Without High-fat/High-caloric Meal: Part 3
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of PF-07202954: Part 3
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-07202954: Part 3
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07202954: Part 1
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: Pharmacokinetic (PK) parameter population included all participants who received at least 1 dose of PF-07202954 and had at least 1 of the PK parameters of interest calculated in Part 1. PK data was not summarized for doses with less than 3 participants as pre-specified in statistical analysis plan; hence, individual values were reported for 'Cohort 2: PF-07202954 100 mg Fasted: Part 1' arm. Treatment groups with same dose and administration were combined as planned.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Cohort 1: PF-07202954 100 mg High Fat/High Calorie Meal: Part 1: Participants were administered a single oral dose of PF-07202954 100 mg with a high fat/ high calorie meal on Day 1 of any treatment period.
Arm/Group | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat/High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 4 | 4 | 9 | 5 | 4 | 5 | 2
Nanogram per milliliter | 23.92 (20) | 55.64 (28) | 226.6 (26) | 774.2 (27) | 2067 (66) | 195.7 (20) | NA (NA) — Data for this arm was not summarized per plan. Individual values for participants were 326 and 290.

14. Secondary Outcome: Time for Cmax (Tmax) of PF-07202954: Part 1
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: PK parameter population included all participants who received at least 1 dose of PF-07202954 and who had at least 1 of the PK parameters of interest calculated in Part 1. Treatment groups with same dose and administration were combined as planned.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 4 | 4 | 9 | 5 | 4 | 5 | 2
Hours | 1.500 [0.500 to 2.00] | 0.7500 [0.500 to 2.00] | 3.000 [0.500 to 4.00] | 1.000 [0.500 to 2.10] | 1.750 [0.500 to 3.00] | 3.000 [0.500 to 4.00] | NA [NA to NA] — It was pre-specified to summarize all PK outcome measures at the group level for 3 or more participants; hence data are not available for this arm.

15. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of PF-07202954: Part 1
Description: AUClast was determined by linear/log trapezoidal method.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: PK parameter population included all participants who received at least 1 dose of PF-07202954 and who had at least 1 of the PK parameters of interest calculated in Part 1. PK data was not summarized for doses with less than 3 participants as pre-specified in the statistical analysis plan; hence, individual values were reported for 'Cohort 2: PF-07202954 100 mg Fasted: Part 1' arm. Treatment groups with same dose and administration were combined as planned.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 4 | 4 | 9 | 5 | 4 | 5 | 2
Nanogram*hour per milliliter | 179.9 (30) | 402.1 (14) | 1905 (27) | 5506 (13) | 13850 (28) | 1834 (28) | NA (NA) — Data for this arm was not summarized per plan. Individual values for participants were 2230 and 2160.

16. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-07202954: Part 1
Description: AUCinf was determined as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable timepoint estimated from the log-linear regression analysis and kel was the terminal phase rate constant. Treatment groups with same dose and administration were combined as planned.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: PK parameter population included all participants who received at least 1 dose of PF-07202954 and who had at least 1 of the PK parameters of interest calculated in Part 1. PK data was not summarized for doses with less than 3 participants as pre-specified in the statistical analysis plan; hence, individual values were reported for 'Cohort 2: PF-07202954 100 mg Fasted: Part 1' arm. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 4 | 4 | 9 | 5 | 4 | 4 | 2
Nanogram*hour per milliliter | 185.6 (29) | 410.1 (14) | 1935 (28) | 5580 (13) | 13980 (28) | 1784 (30) | NA (NA) — Data for this arm was not summarized per plan. Individual values for participants were 2230 and 2180.

17. Secondary Outcome: Terminal Half-life (t1/2) of PF-07202954: Part 1
Description: T1/2 was calculated as loge (2) divided by kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Treatment groups with same dose and administration were combined as planned.
Time Frame: Day 1 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, 48 and 72 hours post-dose)
Population: PK parameter population included all participants who received at least 1 dose of PF-07202954 and who had at least 1 of the PK parameters of interest calculated in Part 1. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
Number analyzed (Participants) | 4 | 4 | 9 | 5 | 4 | 4 | 2
Hours | 5.740 (1.1641) | 5.615 (1.6562) | 11.43 (5.8788) | 10.55 (3.9217) | 14.81 (6.7702) | 15.85 (1.9209) | NA (NA) — It was pre-specified to summarize all PK outcome measures at the group level for 3 or more participants; hence data are not available for this arm.

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07202954 on Day 1, 7 and 14: Part 2
Time Frame: Day 1, 7 and 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Time for Cmax (Tmax) of PF-07202954 on Day 1, 7 and 14: Part 2
Time Frame: Day 1, 7 and 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Groups:
- PF-07202954: Part 2: Participants were planned to receive once daily oral dose of PF-07202954 matching placebo with a standard meal for 14 days.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to Time Tau (AUCtau) of PF-07202954 on Day 1, 7 and 14: Part 2
Description: Area under the concentration curve from time 0 to end of dosing interval (AUCtau).
Time Frame: Day 1, 7 and 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Terminal Half-life (t1/2) of PF-07202954 on Day 14: Part 2
Time Frame: Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Amount of Unchanged Drug Recovered in Urine During Dosing Interval (Aetau) of PF-07202954 on Day 14: Part 2
Description: Aetau was defined as amount of unchanged drug recovered in urine during dosing interval.
Time Frame: Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percent of Dose Recovered in Urine as Unchanged Drug Over Dosing Interval (Aetau%) on Day 14: Part 2
Description: Aetau% was defined as percent of dose recovered in urine as unchanged drug over dosing interval.
Time Frame: Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Renal Clearance (CLr) of PF-07202954 on Day 14: Part 2
Description: Renal clearance was amount of unchanged drug excreted in urine over the dosing interval divided by AUCtau.
Time Frame: Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 8, 10, 12, 14, 16 and 24 hours)
Population: Data was not collected as no participants were enrolled in Part 2 of the study.
Arm/Group | Placebo: Part 2 | PF-07202954: Part 2
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Number of Participants With TEAEs: Part 3
Description: as for outcome 5
Time Frame: Up to maximum of 6 weeks
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Number of Participants With Laboratory Abnormalities Meeting Pre-defined Criteria: Part 3
Description: as for outcome 6
Time Frame: Up to maximum of 6 weeks
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Number of Participants According to Categorization of Vital Signs Data: Part 3
Description: as for outcome 7
Time Frame: Up to maximum of 6 weeks
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Number of Participants According to Categorization of ECG Data: Part 3
Description: as for outcome 8
Time Frame: Up to maximum of 6 weeks
Population: Data was not collected as no participants were enrolled in Part 3 of the study.
Arm/Group | PF-07202954 With High-fat/High-calorie Meal: Part 3 | PF-07202954 Without High-fat/High-calorie Meal: Part 3
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment on Day 1 up to 28 days post last dose of study treatment (maximum up to 10 weeks) for Part 1
Description: Same event may appear as both an AE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Adverse event reported only for Part 1. Since there was no enrolment for Part 2 and 3, hence no safety data collected and reported.
Arm/Group | Cohort 1 and 2: Placebo: Part 1 | Cohort 1: PF-07202954 10 mg: Part 1 | Cohort 2: PF-07202954 30 mg: Part 1 | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 | Cohort 2: PF-07202954 300 mg: Part 1 | Cohort 1: PF-07202954 600 mg: Part 1 | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 | Cohort 2: PF-07202954 100 mg Fasted: Part 1
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4 | 0/4 | 0/9 | 0/5 | 0/4 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 0/4 | 0/9 | 0/5 | 0/4 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 3/11 | 0/4 | 1/4 | 2/9 | 1/5 | 0/4 | 1/5 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and 2: Placebo: Part 1 (N=11) | Cohort 1: PF-07202954 10 mg: Part 1 (N=4) | Cohort 2: PF-07202954 30 mg: Part 1 (N=4) | Cohort 1 and 2: PF-07202954 100 mg Standard Meal: Part 1 (N=9) | Cohort 2: PF-07202954 300 mg: Part 1 (N=5) | Cohort 1: PF-07202954 600 mg: Part 1 (N=4) | Cohort 1: PF-07202954 100 mg High Fat / High Calorie Meal: Part 1 (N=5) | Cohort 2: PF-07202954 100 mg Fasted: Part 1 (N=2)
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Application site irritation (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04857437/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT04857437/SAP_001.pdf